CLINICAL TRIAL: NCT05382169
Title: Prevalence of Mast Cell Activation Syndrome in Patients With Ehlers Danlos Hypermobile Syndrome With Digestive Disorders
Brief Title: Prevalence of Mast Cell Activation Syndrome in Patients With EDS With Digestive Disorders
Acronym: SAMED
Status: Recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P00115
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Ehlers Danlos Hypermobile Syndrome
Keywords: Genetic disease; Collagen abnormality; Nausea; Heartburn; Ehlers Danlos hypermobile syndrome; Mast cell activation syndrome (MCAS); Allergology
MeSH Terms: conditions — Genetic Diseases, Inborn; Nausea; Heartburn; Mast Cell Activation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — basal tryptase blood test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Determine the presence of mast cell activation syndrome — Mast cell activation syndrome will be confirmed if the following three conditions are met (according to Valent et al, 2012) :
  * At least two clinical signs compatible with MAS before the first consultation (V1)
  * Improvement of symptoms on antihistamines within 2 months of initiation of treatment
  * Significant increase in tryptase during crisis
  Mast cell activation syndrome will be possible if :
  * At least two clinical signs consistent with MAS before the first consultation (V1)
  * Improvement of symptoms with antihistamines within 2 months of initiation of treatment
  * No significant increase in tryptase during crisis In all other cases, mast cell activation syndrome is unlikely.

SUMMARY:
The aim of the study is to confirm the association between hypermobile Ehlers Danlos syndrome (hEDS) and mast cell activation syndrome (MCAS) in patients with digestive disorders managed in allergology departments.

ELIGIBILITY:
Inclusion Criteria:

* with hypermobile Ehlers Danlos syndrome
* with digestive disorders
* 14 years of age or older (minimum age for the MOS-SF 36 questionnaire)
* able to answer the questionnaires
* whose participation in a day hospital at Saint Vincent de Paul dedicated to the assessment of "functional digestive pain" is planned
* who do not object to the use of their health data for research purposes

Additional criteria for minors :

- No objection to the use of health data for research purposes by parents/guardians

Exclusion Criteria:

* under guardianship or curatorship
* having taken a long-term high-dose antihistamine treatment (H1 or H2) during the last two months, according to the following thresholds :

  * Desloratadine (>5 mg/jour)
  * Bilastine (>20 mg/jour)
  * Cetirizine (>20 mg/jour)
  * Ebastine (>10 mg/jour)
  * Fexofenadine (>150 mg/jour)
  * Levocetirizine (>5 mg/jour)
  * Loratadine (>10 mg/jour)
  * Exocetiridine (5 mg/jour)
  * Mizolastine (>10 mg/jour)
  * Rupatadine (>10 mg/jour)
  * Polaramine (>10 mg/jour)
  * Oxomemazine (>2 mg/jour)
  * Hydroxyzine (>25 mg/jour)
  * Doxylamine (>15 mg/jour)
  * Cimetidine (>200 mg/jour)
* Patients deprived of liberty, pregnant or nursing women

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with EDSh with digestive disorders
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-28 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of mast cell activation syndrome in patients with hypermobile Ehlers Danlos syndrome with digestive disorders | 2 months
  The presence of mast cell activation syndrome will be described in three modalities : confirmed, possible, and unlikely.
  Mast cell activation syndrome will be confirmed if the following three conditions are met :
  * at least two clinical signs compatible with mast cell activation syndrome (MCAS) before the first consultation (V1)
  * improvement of symptoms with antihistamines within 2 months of initiation of treatment
  * significant increase in tryptase during crisis
  Mast cell activation syndrome will be possible if:
  * at least two clinical signs compatible with MCAS before the first consultation (V1)
  * improvement of symptoms under antihistamine at 2 months of the introduction of the treatment
  * no significant increase in tryptase during crisis In all other cases, mast cell activation syndrome is unlikely.

SECONDARY OUTCOMES:
Frequency of the symptoms after treatment with anti-histamines | 2 months
  Symptoms are those established by Valent et al, 2012. For each clinical sign the patient will rate the frequency of the symptom: more than once a day, once a day, 2 to 6 times a week, once or less a week, never, over the two months prior to visit 1 (V1), and between V1 and the 2-month follow-up visit .
Medical Outcome Study Short-Form 36 (MOS SF-36 ) survey after antihistamine treatment | 2 months
  MOS SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability
Frequency of consumption of analgesics | 2 months
  The frequency of consumption of different analgesics will be studied over the two months preceding V1 and between V1 and V2.
Frequency of intolerance according to particular food consumption | 2 months
  For a given food, at V1 and V2, intolerance will be qualified by the presence of digestive disorders following the consumption of the food among : cow's milk, goat's milk, sheep's milk, fresh cheeses, cow's milk cheese or yogurt, goat's milk cheese or yogurt, sheep's milk cheese or yogurt, wheat/gluten, dry sausage, ham, turkey, chicken, pork, beef, raw egg, cooked egg, smoked fish, canned fish fresh fish, shellfish, mollusks, tomatoes, potatoes, spinach, peas, cabbage, lentils, beans, lemons, oranges, strawberries, raspberries, pineapple, mango, apple, pear, nectarine, peach, banana, kiwi, nuts, peanuts, spices, beers, wines, spirits, other.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette CARON, Md, Principal Investigator — Lille Catholic University
Locations (1):
- Saint-Vincent-de-Paul hospital, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: No